CLINICAL TRIAL: NCT02901691
Title: RHYTHMIC STIMULUS EFFECTS ON NEURONAL OSCILLATORY ACTIVITY AND SPEACHES CAPABILITIES IN DEAF CHILDREN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-31; 2015-A01490-49 (Other: Ansm)
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Children Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deaf children (Experimental)
  Interventions: Other: musical rhythmic stimulation
- healthy volonteer children (Placebo Comparator)
  Interventions: Other: musical rhythmic stimulation

INTERVENTIONS:
Other: musical rhythmic stimulation

SUMMARY:
The deaf children showed deficits in speech processing and temporality. They badly apprehend temporal concepts and perceptions of deficit so the acoustic phenomena marking the time course linguistically. Their prediction capabilities and anticipation multisensory events are thereby affected, thus impacting their ability to adapt to multiple and complex interaction possibilities that arise during a conversation.The project aim it is to measure the impact of a musical rhythmic stimulation of neuronal activity and the temporal prediction capabilities of older deaf children 5 to 8 years and its impact on their language skills in a conversational task. A matched control group of age will be examined for each of the proposed tasks.

We first measure the capacity to anticipate a situation of language interaction. For this purpose, we will use an alternate naming paradigm with a virtual partner, already developed and tested in children with normal hearing. This paradigm approaches the conversational situation while allowing control of the time parameter of speech (speed of trade) and by controlling the bias (temporal) inherent linguistic programming difficulties of children in a spontaneous conversation situations .

Then we will couple behavioral measurements with measurements of eye movements and the electroencephalogram (EEG) in deaf children. For this, we use a dialog observation task already developed for normal hearing children. This task will allow us firstly to analyze the anticipation level of speaking turns by analyzing eye movements (which "precedes" the speaker). Secondly, it will allow us to study the effects of manipulation of the acoustic parameters of auditory evoked potentials (AEP) and the oscillatory activity of the motor system (EEG, mu rhythm and beta). The audiomoteur coupling would seem to be the key point of anticipatory processes and convergence in conversational interaction will also be studied using cortico-cortical coherence techniques to assess the dynamics of connectivity between remote networks (system here auditory and motor system).

ELIGIBILITY:
Inclusion Criteria:

* prélingual paired deaf or implanted cochlear children.

Exclusion Criteria:

* Childreen with other major disabilities and associated disorders.
* Clidren with failure to understand instructions either directly oral or sign language.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Numbers of words and phrases productions in the hearing impaired child. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille; Stéphane ROMAN, MD, Principal Investigator — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No